CLINICAL TRIAL: NCT01595958
Title: CYclosporine A in Non-shockable Out-of-hospital Cardiac Arrest ResUScitation
Brief Title: Cyclosporine A in Cardiac Arrest
Acronym: CYRUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009.571; 2009-015725-37 (EudraCT Number)
Record Dates: First submitted 2012-04-30; First posted 2012-05-10 (Estimated); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Non Shockable Out of Hospital Cardiac Arrest
Keywords: Cardiac arrest; heart arrest; cyclosporine A; post cardiac arrest syndrome; protective agent; multiple organ failure; mitochondrial permeability transition pore; mitochondria; cardio-pulmonary resuscitation; cardioprotection; ischemia reperfusion; postconditioning
MeSH Terms: conditions — Heart Arrest; Post-Cardiac Arrest Syndrome; Multiple Organ Failure | interventions — Cyclosporine; Cardiopulmonary Resuscitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyclosporine A (Experimental): Single intravenous bolus of cyclosporine A (2.5 mg/kg) at the onset of resuscitation
  Interventions: Drug: Cyclosporine A; Procedure: cardio-pulmonary resuscitation
- Control (Active Comparator): usual care of cardiac arrest
  Interventions: Procedure: cardio-pulmonary resuscitation

INTERVENTIONS:
Drug: Cyclosporine A — Single intravenous bolus of cyclosporine A (2.5 mg/kg) at the onset of resuscitation
  Arms: Cyclosporine A
Procedure: cardio-pulmonary resuscitation — usual care of cardiac arrest

SUMMARY:
The investigators hypothesised that cyclosporine A administration at the onset of cardiopulmonary resuscitation, by inhibiting the mitochondrial permeability transition pore, could prevent the post cardiac arrest syndrome and improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Witnessed out-of-hospital cardiac arrest
* Non shockable cardiac rhythm

Exclusion Criteria:

* Evidence of trauma
* Evidence of pregnancy
* Duration of no flow more than 30 minutes
* Rapidly fatal underlying disease
* Allergy to cyclosporin A

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 796 (Actual)
Dates: Start 2010-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Sequential Organ Failure Assessment score (SOFA) | At 24 hours after hospital admission

SECONDARY OUTCOMES:
Hospital admission with return of spontaneous circulation | At 24 hours following admission, at day 28, at hospital discharge (an average time frame of 7 days)
Survival | At 24 hours following admission, at day 28, and at hospital discharge (an average time frame of 7 days)
Good cerebral outcome | At 24 hours following admission, at day 28, and at hospital discharge (an average time frame of 7 days)
  Glasgow Coma Scale and Cerebral Performance Categories
All adverse events | until hospital discharge (an average time frame of 7 days)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent ARGAUD, MD, PhD, Principal Investigator — Groupement Hospitalier Edouard Herriot,69437 Lyon Cedex 03
Locations (1):
- Medical intensive care unit, Edouard Herriot Hospital, Lyon, France

REFERENCES:
- [Result] Argaud L, Cour M, Dubien PY, Giraud F, Jossan C, Riche B, Hernu R, Darmon M, Poncelin Y, Tchenio X, Quenot JP, Freysz M, Kamga C, Beuret P, Usseglio P, Badet M, Anette B, Chaulier K, Alasan E, Sadoune S, Bobbia X, Zeni F, Gueugniaud PY, Robert D, Roy P, Ovize M; CYRUS Study Group. Effect of Cyclosporine in Nonshockable Out-of-Hospital Cardiac Arrest: The CYRUS Randomized Clinical Trial. JAMA Cardiol. 2016 Aug 1;1(5):557-65. doi: 10.1001/jamacardio.2016.1701. PMID 27433815
- [Derived] Madelaine T, Cour M, Roy P, Vivien B, Charpentier J, Dumas F, Deye N, Bonnefoy E, Gueugniaud PY, Coste J, Cariou A, Argaud L. Prediction of Brain Death After Out-of-Hospital Cardiac Arrest: Development and Validation of the Brain Death After Cardiac Arrest Score. Chest. 2021 Jul;160(1):139-147. doi: 10.1016/j.chest.2021.01.056. Epub 2021 Jun 8. PMID 34116828